CLINICAL TRIAL: NCT05423418
Title: A Phase 1 Randomized Study to Evaluate the Safety, Tolerability, and Immunogenicity of Ranging Doses of ALFQ Adjuvant in a Candidate HIV Vaccine Containing A244 and B.65321
Brief Title: Safety, Tolerability, and Immunogenicity of ALFQ in a HIV Vaccine Containing A244 and B.65321 in Healthy Adults
Acronym: RV575
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Military HIV Research Program (Network); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-21-03; RV575 (Other: MHRP); W81XWH1120174 (Other: DAIDS, NIAID, NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus (HIV); AIDS Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A244/B.63521 + 200 μg of ALFQ adjuvant (Active Comparator): Arm 1: An injection containing 300 μg A244 plus 300 μg B.63521 with 200 μg of ALFQ adjuvant will be administered as an IM injection into the deltoid muscle at visits 1, 3, and 5 (corresponding to Day 1, Day 29, and Day 57).
  Interventions: Biological: A244; Biological: B.63521; Biological: 200μg ALFQ
- A244/B.63521 + 100 μg of ALFQ adjuvant (Active Comparator): Arm 2: An injection containing 300 μg A244 plus 300 μg B.63521 with 100 μg of ALFQ adjuvant will be administered as an IM injection into the deltoid muscle at visits 1, 3, and 5 (corresponding to Day 1, Day 29, and Day 57).
  Interventions: Biological: A244; Biological: B.63521; Biological: 100μg ALFQ
- A244/B.63521 + 50 μg of ALFQ adjuvant (Active Comparator): Arm 3: An injection containing 300 μg of A244 plus 300 μg B.63521 with 50 μg of ALFQ adjuvant will be administered as an IM injection into the deltoid muscle at visits 1, 3, and 5 (corresponding to Day 1, Day 29, and Day 57).
  Interventions: Biological: A244; Biological: B.63521; Biological: 50μg ALFQ

INTERVENTIONS:
Biological: A244 — Dose of A244 is 300μg. Vaccine will be administered via IM injection into the same deltoid muscle (same side) for all injections at Month 0 (Day 1), Month 1 (Day 29), and Month 2 (Day 57).
Biological: B.63521 — Dose of B.63521 is 300μg. Vaccine will be administered via IM injection into the same deltoid muscle (same side) for all injections at Month 0 (Day 1), Month 1 (Day 29), and Month 2 (Day 57).
Biological: 50μg ALFQ — Dose of ALFQ is 50μg. Vaccine will be administered via IM injection into the same deltoid muscle (same side) for all injections at Month 0 (Day 1), Month 1 (Day 29), and Month 2 (Day 57).
  Arms: A244/B.63521 + 50 μg of ALFQ adjuvant
Biological: 100μg ALFQ — Dose of ALFQ is 100μg. Vaccine will be administered via IM injection into the same deltoid muscle (same side) for all injections at Month 0 (Day 1), Month 1 (Day 29), and Month 2 (Day 57).
  Arms: A244/B.63521 + 100 μg of ALFQ adjuvant
Biological: 200μg ALFQ — Dose of ALFQ is 200μg. Vaccine will be administered via IM injection into the same deltoid muscle (same side) for all injections at Month 0 (Day 1), Month 1 (Day 29), and Month 2 (Day 57).
  Arms: A244/B.63521 + 200 μg of ALFQ adjuvant

SUMMARY:
This study will evaluate the safety and tolerability (including reactogenicity) of candidate vaccine A244/B.63521 with Army Liposome Formulation (ALF) mixed with the saponin QS-21(Quillaja saponaria-21) (ALFQ) adjuvant. The purpose of this phase I randomized, double-blind clinical trial is to optimize vaccine adjuvant ALFQ dosing by assessing safety, reactogenicity, and immunogenicity. Safety and tolerability will be assessed with both clinical and laboratory monitoring. Sixty human immunodeficiency virus (HIV) negative participants will be enrolled to one of three arms. Vaccinations via intramuscular (IM) injection will occur at months 0, 1, and 2. All participants will receive A244 and B.63521 (300 micrograms of each). In addition, Arm 1 will receive 200 micrograms of ALFQ. Arm 2 will receive 100 micrograms of ALFQ. Arm 3 will receive 50 micrograms of ALFQ.

DETAILED DESCRIPTION:
The purpose of this Phase I randomized, double-blind clinical trial is to optimize ALFQ dosing. Safety will be assessed through the frequency of the overall and specific post-vaccination reactions. Blood will be collected to assess humoral, cell-mediated, and innate immune responses.

Healthy adults not living with HIV who are available for 14 months will be enrolled. A total of 60 participants will be enrolled to one of three arms, each comprised of 20 candidate vaccine recipients. Each arm will receive identical doses of A244 and B.63521 (300 micrograms of each). In addition, Arm 1 will receive 200 micrograms of ALFQ. Arm 2 will receive 100 micrograms of ALFQ. Arm 3 will receive 50 micrograms of ALFQ. The safety, reactogenicity, and immunogenicity will then be compared among the three arms to determine the optimal dose of ALFQ.

All vaccinations will be split into 2 half doses which will both be administered intramuscularly (IM) into the same deltoid muscle. Vaccinations will occur at months 0, 1, and 2. The second vaccination will be administered into the contralateral deltoid at study month 1 compared to the first vaccination at study month 0. The third vaccination at study month 2 will be administered into the same deltoid as the first vaccination at study month 0. Participants will be followed for 12 months following the last study vaccination. Safety and tolerability will be assessed with both clinical and laboratory monitoring. Vaccine- related reactions will be observed and solicited for 30 minutes post-vaccination and with the aid of a diary card and interview of participants during the 14 days post vaccination.

The information gained from the review of the diary card and the interview with the participants will be documented in the clinical study chart. In addition, adverse events (AEs) will be documented at each clinical encounter. AEs will be graded for seriousness, severity, and relationship to the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages 18-55 years (inclusive)
2. Must be at low risk for HIV infection per investigator assessment and using the study risk assessment tool.
3. Able and willing to provide written, informed consent
4. Able and willing to comply with all research requirements, in the opinion of the Investigator
5. Agreement to refrain from blood donation during the course of the study
6. Minimum body weight of 110 pounds (lbs) (50kg)
7. Laboratory Criteria within 30 days before enrollment:

   1. Hemoglobin ≥ 12.0 g/dL for women; ≥ 12.5 g/dL for men
   2. White Blood Cell count = 3,500-10,800 cells/mm3
   3. Platelets ≥140,000/mm3 and ≤ 450,000/mm3
   4. Alanine aminotransferase (ALT; SGPT) <1.25 x Upper Limit of Normal (ULN)
   5. Serum creatinine ≤ 1.25 x institutional upper limit of the reference range
   6. Negative HIV testing (HIV Ab / antigen 4th generation screen with reflex confirmatory RNA testing)
   7. Negative HBsAg and hepatitis C antibody testing Note: As above, Grade 1 lab abnormalities detected on screening may be repeated at PI discretion. Persistent Grade 1 abnormalities that are felt to represent the non-pathologic baseline for the subject will be documented before a subject is enrolled in the trial and are allowable per discretion of the PI.
8. Birth control requirements:

   All participants assigned female at birth must meet one of the following 2 criteria:
   1. No reproductive potential due to post-menopausal status (12 months of natural [spontaneous] amenorrhea) or hysterectomy, bilateral oophorectomy, or tubal ligation
   2. People of childbearing potential should agree to practice highly effective contraception at least 30 days before enrollment and through 3 months post-last vaccination, using one of the following methods: condoms (male or female) with spermicide; diaphragm, or cervical cap with spermicide; intrauterine device; contraceptive pills, patch, injection, intravaginal ring or other FDA-approved contraceptive method; male partner has previously undergone a vasectomy; abstinence
   3. All participants are encouraged to engage in safe sex practices to prevent HIV acquisition
9. For all participants assigned female at birth, except those with a history of hysterectomy or bilateral oophorectomy, a negative β-human chorionic gonadotropin (HCG) pregnancy test (urine) on the day of enrollment and each vaccination day is required. Because tubal ligations have a failure rate that is not insignificant, and because 12 months of spontaneous amenorrhea can be a result of polycystic ovarian syndrome and does not completely preclude pregnancy, a negative β- HCG pregnancy test at enrollment and on each vaccination day is also required for participants assigned female at birth with a history of either of these).
10. No plans to travel outside the Washington DC metro area (DC, Maryland, and Virginia) that would prevent compliance with planned study visits
11. Test of Understanding (TOU) (minimum passing score of 80% with 2 attempts permitted)

Exclusion Criteria:

1. Receipt of any investigational HIV vaccine or investigational adjuvant
2. Received an investigational product in the 30 days before enrollment, or planned to receive during the study period. This does not include products with emergency use authorization.
3. Concurrent participation in another clinical research study
4. Any serious medical illness or condition
5. Receipt of immunoglobulins or blood products within 3 months before enrollment
6. Any history of anaphylaxis or allergy to study product
7. History of sickle cell trait or disease
8. Pregnancy, lactation, or intention to become pregnant during the study
9. History of active/recent cancer still within treatment or active surveillance follow-up (except basal cell carcinoma of the skin and cervical carcinoma in situ). Treated/resolved cancers with no likelihood of recurrence may be deemed acceptable at Principal Investigator (PI) discretion.
10. History of autoimmune disease
11. History of Potentially Immune-Mediated Medical Conditions (PIMMCs)
12. Suspected or known current alcohol or drug abuse as defined by an alcohol intake of greater than 3 drinks a day on average for a man, and greater than 2 drinks a day on average for a woman
13. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to give informed consent, participate in the study, or impair interpretation of the study data, in the opinion of the Investigator
14. History of splenectomy
15. History of confirmed or suspected immunodeficiency
16. History of hereditary angioedema (HAE) acquired angioedema (AAE), or idiopathic forms of angioedema
17. History of asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years
18. History of diabetes mellitus (type I or II), with the exception of gestational diabetes
19. History of thyroid disease (except for well controlled hypothyroidism)
20. History of idiopathic urticaria within the past year
21. History of hypertension that is not well controlled by medication or that is persistently greater than 140/95 at screening
22. History of bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
23. History of chronic or active neurologic disease to include seizure disorder and chronic migraine headaches. Exceptions are: i) childhood febrile seizures, or ii) seizures secondary to alcohol withdrawal more than 3 years ago
24. Subjects receiving any of the following substances:

    1. Systemic immunosuppressive medications or cytotoxic medications within 12 weeks before enrollment [with the exception of a short course of corticosteroids (≤ 14 days duration or a single injection) for a self-limited condition at least 2 weeks before enrollment; inhaled, intranasal or topical steroids are not considered exclusionary
    2. Treatment with known immunomodulators including allergy immunotherapy (other than nonsteroidal anti-inflammatory drugs [NSAIDs] or stable maintenance immunotherapy (doses not in the process of being increased), at the discretion of the Protocol Safety Review Team (PSRT)) for any reason
    3. Live attenuated vaccines within 30 days before initial study vaccine administration
    4. Medically indicated subunit, messenger ribonucleic acid (mRNA), or killed vaccines, e.g., influenza, pneumococcal, vaccines with Quillaja saponaria-21 (QS-21) as an adjuvant, or allergy treatment with antigen injections, planned for administration 14 days before or after study vaccine administration
25. History of arthritis diagnosis other than osteoarthritis
26. History of other diagnosed rheumatoid disorders
27. Has an acute illness or temperature ≥38.0 degrees Celsius (C)/100.4 degrees Fahrenheit (F) on any study injection day or within 48 hours of planned study injection.

Note: Participants will not be excluded from further consideration for enrollment and study injections. Volunteers with fever or an acute illness on the day of study injection or in the 2 days before the study injection may be re-assessed by a study physician for resolution of the condition and enrolled and receive the study injection so long as the injection is within allowable windows. Military personnel will be excluded from participation in this study, regardless of leave status due to the potential for a false-positive HIV test result on mandatory HIV testing. This could have adverse effects on deployment status.

Final evaluation of eligibility will be based on the medical judgment of the investigator based on his/her medical and research experience.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), Serious Adverse Events (SAE), Adverse Events of Special Interest (AESI), and unsolicited AEs | Days 0 to 393
  The number of participants with AEs, SAEs, AESIs, and unsolicited AEs on Day 0 through Day 337 as assessed by the Division of AIDS (DAIDS) grading scale and possible attribution to Investigational Product. The number of participants with medically attended AE will be followed until Day 393.
Number of Participants with Local and Systemic Reactions | Days 0 to 14 post vaccination
  Post-vaccination reactions, including redness/erythema, induration, pain/tenderness, itching, warmth, fever, chills, myalgia, arthralgia, headache, nausea, fatigue, rash, and dizziness, will be assessed and recorded on diary cards on Days 0 through 14.

SECONDARY OUTCOMES:
Number of Participants with HIV-specific Binding Antibodies | Day 0 to 336
  Vaccine-induced humoral immune responses will be assessed by HIV-specific binding antibody assays, HIV-specific neutralizing antibody assays, and non-neutralizing antibody function assays. HIV-specific cell-mediated responses will be assessed by intracellular cytokine staining, cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) T cell proliferation, and related assays. Innate immune responses and genetic responses will be assessed with flow cytometric panels, DNA microarrays, and RNA sequencing. Blood draws to complete assessments will be obtained at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Cebula, MD, Principal Investigator — Research Physician at U.S. Military HIV Research Program
Locations (1):
- Walter Reed Army Institute of Research, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam SM, Liao HX, Tomaras GD, Bonsignori M, Tsao CY, Hwang KK, Chen H, Lloyd KE, Bowman C, Sutherland L, Jeffries TL Jr, Kozink DM, Stewart S, Anasti K, Jaeger FH, Parks R, Yates NL, Overman RG, Sinangil F, Berman PW, Pitisuttithum P, Kaewkungwal J, Nitayaphan S, Karasavva N, Rerks-Ngarm S, Kim JH, Michael NL, Zolla-Pazner S, Santra S, Letvin NL, Harrison SC, Haynes BF. Antigenicity and immunogenicity of RV144 vaccine AIDSVAX clade E envelope immunogen is enhanced by a gp120 N-terminal deletion. J Virol. 2013 Feb;87(3):1554-68. doi: 10.1128/JVI.00718-12. Epub 2012 Nov 21. PMID 23175357
- [Background] Cawlfield A, Genito CJ, Beck Z, Bergmann-Leitner ES, Bitzer AA, Soto K, Zou X, Hadiwidjojo SH, Gerbasi RV, Mullins AB, Noe A, Waters NC, Alving CR, Matyas GR, Dutta S. Safety, toxicity and immunogenicity of a malaria vaccine based on the circumsporozoite protein (FMP013) with the adjuvant army liposome formulation containing QS21 (ALFQ). Vaccine. 2019 Jun 27;37(29):3793-3803. doi: 10.1016/j.vaccine.2019.05.059. Epub 2019 May 28. PMID 31151801
- [Background] Gray GE, Bekker LG, Laher F, Malahleha M, Allen M, Moodie Z, Grunenberg N, Huang Y, Grove D, Prigmore B, Kee JJ, Benkeser D, Hural J, Innes C, Lazarus E, Meintjes G, Naicker N, Kalonji D, Nchabeleng M, Sebe M, Singh N, Kotze P, Kassim S, Dubula T, Naicker V, Brumskine W, Ncayiya CN, Ward AM, Garrett N, Kistnasami G, Gaffoor Z, Selepe P, Makhoba PB, Mathebula MP, Mda P, Adonis T, Mapetla KS, Modibedi B, Philip T, Kobane G, Bentley C, Ramirez S, Takuva S, Jones M, Sikhosana M, Atujuna M, Andrasik M, Hejazi NS, Puren A, Wiesner L, Phogat S, Diaz Granados C, Koutsoukos M, Van Der Meeren O, Barnett SW, Kanesa-Thasan N, Kublin JG, McElrath MJ, Gilbert PB, Janes H, Corey L; HVTN 702 Study Team. Vaccine Efficacy of ALVAC-HIV and Bivalent Subtype C gp120-MF59 in Adults. N Engl J Med. 2021 Mar 25;384(12):1089-1100. doi: 10.1056/NEJMoa2031499. PMID 33761206
- [Background] Gray GE, Allen M, Moodie Z, Churchyard G, Bekker LG, Nchabeleng M, Mlisana K, Metch B, de Bruyn G, Latka MH, Roux S, Mathebula M, Naicker N, Ducar C, Carter DK, Puren A, Eaton N, McElrath MJ, Robertson M, Corey L, Kublin JG; HVTN 503/Phambili study team. Safety and efficacy of the HVTN 503/Phambili study of a clade-B-based HIV-1 vaccine in South Africa: a double-blind, randomised, placebo-controlled test-of-concept phase 2b study. Lancet Infect Dis. 2011 Jul;11(7):507-15. doi: 10.1016/S1473-3099(11)70098-6. Epub 2011 May 11. PMID 21570355
- [Background] Liao HX, Tsao CY, Alam SM, Muldoon M, Vandergrift N, Ma BJ, Lu X, Sutherland LL, Scearce RM, Bowman C, Parks R, Chen H, Blinn JH, Lapedes A, Watson S, Xia SM, Foulger A, Hahn BH, Shaw GM, Swanstrom R, Montefiori DC, Gao F, Haynes BF, Korber B. Antigenicity and immunogenicity of transmitted/founder, consensus, and chronic envelope glycoproteins of human immunodeficiency virus type 1. J Virol. 2013 Apr;87(8):4185-201. doi: 10.1128/JVI.02297-12. Epub 2013 Jan 30. PMID 23365441
- [Background] Pitisuttithum P, Nitayaphan S, Chariyalertsak S, Kaewkungwal J, Dawson P, Dhitavat J, Phonrat B, Akapirat S, Karasavvas N, Wieczorek L, Polonis V, Eller MA, Pegu P, Kim D, Schuetz A, Jongrakthaitae S, Zhou Y, Sinangil F, Phogat S, Diazgranados CA, Tartaglia J, Heger E, Smith K, Michael NL, Excler JL, Robb ML, Kim JH, O'Connell RJ, Vasan S; RV306 study group. Late boosting of the RV144 regimen with AIDSVAX B/E and ALVAC-HIV in HIV-uninfected Thai volunteers: a double-blind, randomised controlled trial. Lancet HIV. 2020 Apr;7(4):e238-e248. doi: 10.1016/S2352-3018(19)30406-0. Epub 2020 Feb 6. PMID 32035516

DOCUMENTS (3):
  • Study Protocol (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT05423418/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT05423418/SAP_001.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT05423418/ICF_002.pdf